CLINICAL TRIAL: NCT03101072
Title: The PIRATE PROJECT: a Point-of-care, Informatics-based Randomized Controlled Trial for Decreasing Over-utilization of Antibiotic ThErapy in Gram-negative Bacteremia
Brief Title: Antibiotic Durations for Gram-negative Bacteremia
Acronym: PIRATE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Geneva, Switzerland (Other)
Collaborators: Centre Hospitalier Universitaire Vaudois (Other); Cantonal Hospital of St. Gallen (Other)
Responsible Party: Principal Investigator, Angela HUTTNER, Principal Investigator, University of Geneva, Switzerland
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2017-00108
Record Dates: First submitted 2017-03-29; First posted 2017-04-04 (Actual); Last update posted 2019-11-19 (Actual); Status verified 2019-11

CONDITIONS: Bacteraemia Caused by Gram-Negative Bacteria
Keywords: Gram-negative bacteremia; antibiotic durations; point-of-care randomization

STUDY DESIGN:
Intervention Model Description: With day 1 defined as the first day of appropriate (microbiologically efficacious) antibacterial therapy, patients will be randomized 1:1:1 on day 5 (±1) to one of the following three arms:
  * "Fixed long" antibiotic course of 14 days (control arm)
  * "Fixed short" antibiotic course of 7 days (first intervention arm)
  * "Individualized" antibiotic course (second intervention arm): • Starting on day 5, therapy will be discontinued after the patient has been afebrile for 48 hours and the CRP level has decreased from its peak by at least 75% In all arms, the choice and mode of administration (IV vs. PO) of antibiotic(s) will be left to the patient's attending physician and consulting infectious disease specialist and thus will follow usual standards of care.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants, their care providers, and study investigators having contact with participants & their providers will be blinded until the antibiotic therapy is discontinued. Outcomes assessors and data analysts will be fully blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- "Fixed long" antibiotic course (Active Comparator): Patients randomized to this group will receive a "fixed long" antibiotic course of 14 days.
  Interventions: Other: "Fixed long" antibiotic course of 14 days
- "Fixed short" antibiotic course (Experimental): Patients randomized to this group will receive a "fixed short" antibiotic course of 7 days.
  Interventions: Other: "Fixed short" antibiotic course of 7 days
- "Individualized" antibiotic course (Experimental): "Individualized" antibiotic course: starting on day 5, therapy will be discontinued after the patient has been afebrile for 48 hours and the CRP level has decreased from its peak by at least 75%
  Interventions: Other: "Individualized duration" of antibiotic therapy

INTERVENTIONS:
Other: "Fixed long" antibiotic course of 14 days — Only the duration of antibiotic therapy will be investigated in this study. (In all arms, the choice and mode of administration (IV vs. PO) of antibiotic(s) will be left to the patient's attending physician and consulting infectious disease specialist and thus will follow usual standards of care.)
  Arms: "Fixed long" antibiotic course
Other: "Fixed short" antibiotic course of 7 days — Only the duration of antibiotic therapy will be investigated in this study. (In all arms, the choice and mode of administration (IV vs. PO) of antibiotic(s) will be left to the patient's attending physician and consulting infectious disease specialist and thus will follow usual standards of care.)
  Arms: "Fixed short" antibiotic course
Other: "Individualized duration" of antibiotic therapy — Only the duration of antibiotic therapy will be investigated in this study. (In all arms, the choice and mode of administration (IV vs. PO) of antibiotic(s) will be left to the patient's attending physician and consulting infectious disease specialist and thus will follow usual standards of care.)
  Arms: "Individualized" antibiotic course

SUMMARY:
Gram-negative bacteremia (GNB) is a frequent hospital & community-acquired infection, yet there is as yet no evidence from randomized studies on the optimal duration of antibiotic therapy. This point-of-care, multicenter randomized controlled non-inferiority trial will randomize 500 patients with GNB on day 5 of appropriate antibiotic therapy to either (1) a total of 7 days of antibiotic therapy, (2) a total of 14 days of antibiotic therapy, or (3) an individualized duration of antibiotic therapy (guided by the patient's clinical course & C-reactive protein levels). The primary outcome is the incidence of clinical failure at day 30.

DETAILED DESCRIPTION:
Antibiotic resistance continues to grow and is now considered to be one of the most serious global threats of the 21st century. The key driver of resistance is antibiotic overuse; long antibiotic courses select for resistance among the trillions of bacteria hosted by the human body. There is as yet no evidence from randomized studies on its optimal duration of antibiotic therapy. Traditionally, guidelines have somewhat arbitrarily recommended long courses of two weeks, even though patients with no structural complications may recover after only five days of therapy. Evidence is mounting that longer courses leave patients with multi-resistant organisms. Indeed, given rising concerns over resistance, many physicians have reduced antibiotic durations for GNB to 7 days with no apparent untoward consequences.

This point-of-care, multicenter randomized controlled non-inferiority trial will randomize 500 patients with GNB on day 5 of appropriate antibiotic therapy to either (1) a total of 7 days of antibiotic therapy, (2) a total of 14 days of antibiotic therapy, or (3) an individualized duration of antibiotic therapy (guided by the patient's clinical course & C-reactive protein levels). The primary outcome is the incidence of clinical failure at day 30. Patients will be followed through day 90; secondary outcomes will include the incidence of clinical failure on days 60 and 90, the total number of antibiotic days, the incidence of antibiotic-related adverse events (including Clostridium difficile infection), the emergence of bacterial resistance, length of hospital stay. Cost-effectiveness/health-economic analyses will also be performed.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Presence of Gram-negative bacteria in at least one blood culture bottle
3. Treatment with a microbiologically efficacious antibiotic

Exclusion Criteria:

1. Immunosuppression (including HIV infection with CD4 cell count ≤500/µl, hematopoietic stem-cell transplantation in the first month after transplantation and at any time before engraftment, neutropenia in the 48 hours prior to randomization, receipt of high-dose steroids [>40 mg prednisone or its equivalent] daily for > 2 weeks) in the two weeks prior to randomization
2. GNB due to the following complicated infections:

   * Endocarditis or other endovascular infection without a removable focus
   * Necrotizing fasciitis
   * Osteomyelitis or septic arthritis
   * Confirmed prostatitis
   * Undrainable abscess or other unresolved sources requiring surgical intervention (e.g., cholecystitis) at the time of enrollment
   * Central nervous system infections
   * Empyema
3. GNB due to non-fermenting bacilli (Acinetobacter spp., Burkholderia spp., Pseudomonas spp.), Brucella spp., Fusobacterium spp., or polymicrobial growth with Gram-positive organisms
4. Fever (≥38º C) or hemodynamic instability in the 24h prior to recruitment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 504 (Actual)
Dates: Start 2017-04-27 (Actual); Primary Completion 2019-06-11 (Actual); Study Completion 2019-08-26 (Actual)

PRIMARY OUTCOMES:
Incidence of clinical failure in all arms | day 30 (with day 1 being the first day of microbiologically efficacious antibiotic therapy)
  Clinical failure is defined by the presence of at least one of the following:
  * Relapse: a recurrent bacteremia due to the same bacterium occurring from the day of treatment cessation and until day 30
  * Local suppurative complication that was not present/apparent at infection onset (e.g., renal abscess in pyelonephritis, empyema in pneumonia)
  * Distant complications of the initial infection, defined by growth of the same bacterium causing the initial bacteremia (as determined by antibiotic susceptibility profiling)
  * The restarting of Gram-negative-directed antibiotic therapy after its initial discontinuation due to clinical worsening suspected to be due to the initial infecting organism and for which there is no alternate diagnosis/pathogen suspected
  * Death due to any cause through day 30

SECONDARY OUTCOMES:
Incidence of clinical failure in all arms | day 60
  Clinical failure is defined by the presence of at least one of the following:
  * Relapse: a recurrent bacteremia due to the same bacterium occurring from the day of treatment cessation and until day 30
  * Local suppurative complication that was not present/apparent at infection onset (e.g., renal abscess in pyelonephritis, empyema in pneumonia)
  * Distant complications of the initial infection, defined by growth of the same bacterium causing the initial bacteremia (as determined by antibiotic susceptibility profiling)
  * The restarting of Gram-negative-directed antibiotic therapy after its initial discontinuation due to clinical worsening suspected to be due to the initial infecting organism and for which there is no alternate diagnosis/pathogen suspected
  * Death due to any cause through day 30
Incidence of clinical failure in all arms | day 90
  Clinical failure is defined by the presence of at least one of the following:
  * Relapse: a recurrent bacteremia due to the same bacterium occurring from the day of treatment cessation and until day 30
  * Local suppurative complication that was not present/apparent at infection onset (e.g., renal abscess in pyelonephritis, empyema in pneumonia)
  * Distant complications of the initial infection, defined by growth of the same bacterium causing the initial bacteremia (as determined by antibiotic susceptibility profiling)
  * The restarting of Gram-negative-directed antibiotic therapy after its initial discontinuation due to clinical worsening suspected to be due to the initial infecting organism and for which there is no alternate diagnosis/pathogen suspected
  * Death due to any cause through day 30
Incidence of all-cause mortality in all arms | day 90
  incidence of all-cause mortality
Incidence of Clostridium difficile infection in all arms | day 90
  incidence of symptomatic C. difficile infection in all arms
Incidence of emergence of resistance to the study antibiotic in all arms | day 90
  The incidence of emergence of resistance in micro-organisms recovered in clinical specimens (whether colonizers or etiologic agents of the gram-negative bacteremia) in all arms

CONTACTS AND LOCATIONS:
Overall Officials: Angela Huttner, MD, Principal Investigator — University of Geneva
Locations (3):
- Switzerland (3):
  - Cantonal Hospital St Gallen, Sankt Gallen, Canton of St. Gallen
  - Lausanne University Hospital, Lausanne, Canton of Vaud
  - Geneva University Hospitals, Geneva

IPD SHARING:
Plan to Share IPD: No
(There is no plan to share IPD.)

REFERENCES:
- [Derived] von Dach E, Albrich WC, Brunel AS, Prendki V, Cuvelier C, Flury D, Gayet-Ageron A, Huttner B, Kohler P, Lemmenmeier E, McCallin S, Rossel A, Harbarth S, Kaiser L, Bochud PY, Huttner A. Effect of C-Reactive Protein-Guided Antibiotic Treatment Duration, 7-Day Treatment, or 14-Day Treatment on 30-Day Clinical Failure Rate in Patients With Uncomplicated Gram-Negative Bacteremia: A Randomized Clinical Trial. JAMA. 2020 Jun 2;323(21):2160-2169. doi: 10.1001/jama.2020.6348. PMID 32484534
- [Derived] Huttner A, Albrich WC, Bochud PY, Gayet-Ageron A, Rossel A, Dach EV, Harbarth S, Kaiser L. PIRATE project: point-of-care, informatics-based randomised controlled trial for decreasing overuse of antibiotic therapy in Gram-negative bacteraemia. BMJ Open. 2017 Jul 13;7(7):e017996. doi: 10.1136/bmjopen-2017-017996. PMID 28710229